CLINICAL TRIAL: NCT04901091
Title: Study of the Immediate and Long-term Outcomes of the Disease in Patients With Left Ventricular Aneurysm Complicated and Uncomplicated by Thrombosis After Transmural Myocardial Infarction, According to the Hospital Registry
Brief Title: Study of the Immediate and Long-term Outcomes of the Disease in Patients With Left Ventricular Aneurysm Complicated and Uncomplicated by Thrombosis After Transmural Myocardial Infarction, According to the Hospital Registry: SIBYL
Acronym: SIBYL
Status: Completed | Type: Observational
Sponsor: National Medical Research Center for Therapy and Preventive Medicine (Other Government)
Collaborators: N.V. Sklifosovsky Research Institute for Emergency Medicine of the Moscow Healthcare Department (Unknown)
Responsible Party: Sponsor
Other Study IDs: 01-05-21
Record Dates: First submitted 2021-05-14; First posted 2021-05-25 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Myocardial Infarction
Keywords: left ventricular aneurysm, transmural myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- study group№ 1: patients who have left ventricular aneurysm without thrombosis
  Interventions: Other: Not Provided
- study group№ 2: patients who have left ventricular aneurysm with thrombosis
  Interventions: Other: Not Provided
- control group: patients who have not left ventricular aneurysm
  Interventions: Other: Not Provided

INTERVENTIONS:
Other: Not Provided — Not Provided

SUMMARY:
A prospective non-interventional study aimed to evaluate the immediate and long-term outcomes in patients with left ventricular aneurysm after transmural myocardial infarction.

A registry of patients with transmural myocardial infarction admitted to the Emergency Department of Cardiology will be created. The registry will include all consecutive hospitalized patients from from January 1, 2021 to December 31, 2021 who meet the inclusion criteria Based on this registry, patients will be divided into groups : patients with left ventricular aneurysm and patients without aneurysm, patients with left ventricular thrombosis and patients without thrombosis.

Patients will be contacted in 3 and 12 months. Surviving patients will be invited to appointment for an ECG, echocardiography and survey. The cardiovascular events during this period will be recorded.

The factors determining the prognosis of patients and their concomitant diseases, immediate and long-term prognoses, therapeutic measures and drug therapy at the hospital and outpatient stages, and patients ' adherence to therapy will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women who had acute transmural myocardial infarction and who were hospitalized to the Emergency Cardiology Department of the N. V. Sklifosovsky Research Institute of Emergency Medicine from January 1, 2021 to December 31, 2021
2. Patients from 18 to 85 years of age
3. Patients who live in Moscow and Moscow region
4. Patients who signed the consent to participate in the study and processing of personal data.

Exclusion Criteria:

1. Patients who refused to come for a second appointment or answer the questionnaire questions
2. Patients who had repeated myocardial infarction
3. Non-compliance with inclusion criteria

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with transmural myocardial infarction admitted to the Emergency Department of Cardiology
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 12 months
  Patients with a fatal outcome will be identified. We will contact the relatives of the deceased patients to clarify the date of death.

SECONDARY OUTCOMES:
Cumulative number cardiovascular events | 12 months
  Cardiovascular event is defined on of the following repeated myocardial infarctions, brain strokes, PCI, CABG, pulmonary embolism.
Assessment of adherence | baseline, 3 months, 12 months
  To assess adherence to the recommended therapy at enrollment and during the first and second visits, the original questionnaire "The Scale of Adherence of the National Society for Evidence-based Pharmacotherapy" will be used. The commitment scale has two modifications to assess potential and initial actual commitment. The questionnaire can be used both to assess overall adherence to drug therapy and to diagnose adherence to a specific drug.
  The maximum number of points on the scale is 4 points. The minimum number of points on the scale is 0 points. 4 points means complete non-adherence. 0 points means full commitment.

CONTACTS AND LOCATIONS:
Locations (1):
- N.V. Sklifosovsky Research Institute for Emergency Medicine of the Moscow Healthcare Department, Moscow, Russia